CLINICAL TRIAL: NCT02146898
Title: The Severity Of Hypotension Comparing Three Positions During Spinal Anesthesia For Cesarean Delivery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Phillip Hess, Chief of Obstetric Anesthesia, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013P000171
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Last update posted 2017-01-04 (Estimated); Status verified 2017-01

CONDITIONS: Hypotension
Keywords: spinal anesthesia; hypotension; pregnancy
MeSH Terms: conditions — Hypotension | interventions — Patient Positioning

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lateral (Active Comparator): patient placed in the lateral postion for spinal anesthesia
  Interventions: Other: Position
- Sitting (Active Comparator): patient placed in the sitting position for spinal anestheisa, then supine
  Interventions: Other: Position
- Recline (Active Comparator): patient placed in the sitting position for spinal anesthesia administration. After spinal placed, the patient turned to a 30-degree upperbody tilt, followed by a slow recline to supine over 5 minutes
  Interventions: Other: Position

INTERVENTIONS:
Other: Position

SUMMARY:
The investigators intend to study the impact of patient positioning on the changes in blood pressure after spinal anesthesia for cesarean delivery. The investigators hypothesized that the changes in blood pressure relate to the speed with which the spinal medication rises. By slowing the rise of spinal anesthesia, the investigators believe that the incidence and severity of hypotension might be reduced.

DETAILED DESCRIPTION:
Spinal anesthesia is the most commonly used anesthetic for cesarean delivery. In part, this is due to the ease of administration, reliability and low rates of adverse effects. Additionally, the avoidance of general anesthesia allows the parturient to participate in the birth experience, despite being in surgery.

Although hyperbaric local anesthetic solutions have a remarkable record of safety, their use is not totally without risk. The side effects of spinal anesthesia are well described, but most notably include hypotension (low blood pressure). Spinal hypotension is primarily due to the vasodilatory effects of local anesthetics, and would occur in virtually all women if not prevented or treated.

The incidence of hypotension in both the literature and in clinical practice ranges from 30% to 50% of all patients. Recent literature using a continuous, non-invasive blood pressure monitor suggests that hypotension occurs with greater frequency and may be associated with a higher incidence of adverse effects to either mother or fetus. The incidence and degree of hypotension have been associated with fetal acidosis, which is a sign of either poor perfusion of the placental bed, or increased metabolism due to the blood pressure medications.

The most effective treatment for spinal hypotension is uterine displacement using a hip wedge; the use of a hip wedge after spinal anesthesia is a standard of care. Other treatment, including fluid administration of either crystalloid or colloid, are either partially effective, clinical impractical, or result in administering large doses of medications that may have negative effects on the fetus.

Epidural anesthesia is associated with a reduction in the incidence and severity of hypotension compared with spinal anesthesia. This is believed to be due to the slower onset of sympathetic blockade with epidural anesthesia; this slow onset allows the physiologic compensation to changes in blood pressure. Unfortunately, the slower onset and lower reliability of epidural anesthesia prevents routine use in clinical practice for cesarean delivery.

The investigators hypothesize that the position patients are in during spinal placement might play a role in the severity of maternal hypotension. Interestingly, very few studies have investigated this posibility. Gori, et al. (1) studied influence of seated versus lateral positioning for spinal placement in Cesarean section. They found no significant differences in onset times, Bromage score for motor block, recovery dynamics, and use of ephedrine in two different positions; however, they did not compare the incidence and severity of spinal hypotension. Yun, et al. (2) found that the severity and duration of hypotension were greater when hyperbaric bupivacaine and fentanyl were induced in the sitting position compared to lateral.

Of notice, in all these studies, the authors focused on the immediate positions when the spinal mediation was injected; none has examined the effect of positioning after injection during phase when spinal anesthesia is rising.

Density differences between intrathecal injectate and CSF may explain the observed postural differences in extent of sensory block. Thus, the height of spinal anesthesia blockade could be affected by patient positioning during and after spinal injection. A small incline in positioning immediately after spinal injection may slow the rise of spinal blockade without affecting the duration of spinal anesthesia. In the current protocol, the investigators hypothesize that by slowing the rise of spinal anesthesia, the investigators might reduce the severity of hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Term gestation
* Scheduled cesarean delivery
* Spinal anesthesia for delivery

Exclusion Criteria:

* Significant fetal concerns
* Polyhydramnios
* Macrosomia
* Morbid obesity (BMI >40)
* Chronic hypertension
* Gestational hypertension
* Preeclampsia
* Type 1 diabetes
* Contraindications to spinal anesthesia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2013-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
change in blood pressure | 20 minutes
  percentage change in blood pressure after spinal anesthesia

SECONDARY OUTCOMES:
IV fluid administration | 20 minutes
  Difference in IV fluid requirements

OTHER OUTCOMES:
IV pressor requirements | 20 minutes
  Requirements for IV administration of vasopressors

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Isreal Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No